CLINICAL TRIAL: NCT03972098
Title: Uromodulin Levels in Rheumatoid Arthritis
Brief Title: Uromodulin in Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: neval aksoy (Other)
Responsible Party: Sponsor-Investigator, neval aksoy, Medical Doctor, Head of Urine Laboratory Department, Istanbul Saglik Bilimleri University
Organization: Istanbul Saglik Bilimleri University (Other)
Other Study IDs: Gaziosmanpasa Hospital
Record Dates: First submitted 2019-05-04; First posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Rheumatoid Arthritis
Keywords: uromodulin
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ra patients: The diagnosis of RA was based on the criteria developed by the American College of Rheumatology and European League Against Rheumatism (ACR/EULAR) in 2010 [8]. A drug history was obtained from every patient. All non-steroidal anti-inflammatory medications and disease-modifying antirheumatic drugs prescribed during the year before enrollment in the study were recorded. criteria included systemic diseases (renal failure, hepatic insufficiency, diabetes mellitus, other collagen vascular diseases, history of smoking and consumption of alcohol.In order to eliminate the possibility of any systemic disease therefore we choose that our control group as young.
- healthy control: healthy person, similar population

SUMMARY:
The aim of the present study was to evaluate the levels of uromodulin in rheumatoid arthritis (RA) and to investigate whether it was correlated with baseline clinical characteristics. In addition CKD epi,MDRD,urine microalbuminuria,pH,serum urea, creatinine,CRP (C-Reactive protein) were measured.The participants consist of ; %68 patients,% 32 control group.

DETAILED DESCRIPTION:
Uromodulin, also known as Tamm-Horsfall protein, is a protein abundantly excreted in the urine in healthy individuals. It is synthesized in the thick ascending limb of Henle (TALH) and the early distal convoluted tubule. Its biologic function is still obscure; however, some experimental studies indicated that it might serve as an important urinary defense factor against bacterial colonization and stone formation.

There are controversial publications on the frequencies of urinary tract infections and nephrolithiasis in patients with mutations of uromodulin gene. Deposition of mutated uromodulin in the urinary system may lead to tubular cell dysfunction and apoptosis. These alterations may subsequently cause tubular atrophy and interstitial fibrosis . Moreover, the release of abnormal uromodulin after apoptosis through basolateral secretion may elicit an immune response which may give rise to an immune-mediated tubulointerstitial nephritis .

Uromodulin can activate the other components of the immune system and may modulate the inflammatory and immune responses through different mechanisms .

Experimental studies yielded that uromodulin negative mice displayed splenomegaly with infiltration of white pulp by macrophages and increased levels of TNF-α and interleukin-1 . Rheumatoid arthritis is a systemic autoimmune condition that may eventually result in the joint damage, disability and premature mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients who diagnosed of rheumatoid arthritis as criteria of ACR/EULAR 2010.
* All patients age range is 18-80 years.

Exclusion Criteria :

* Renal failure
* Hepatic insufficiency
* Diabetes mellitus
* Other collagen vascular diseases,
* History of smoking and consumption of alcohol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A drug history was obtained from every patient. All non-steroidal anti-inflammatory medications and disease-modifying antirheumatic drugs prescribed during the year before enrollment in the study were recorded.
  In order to eliminate the possibility of any systemic disease therefore we choose that our control group as young
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Patients with rheumatoid arthritis | 1 day
  The diagnosis of RA was based on the criteria the American College of Rheumatology and European League Against Rheumatism (ACR/EULAR) in 2010.
  Patients selected
  1. have at least 1 joint with definite clinical synovitis (swelling)
  2. with the synovitis not better explained by another disease Classification criteria for RA (score-based algorithm: add score of categories A-D; a score of >6/10 is needed for classification of a patient as having definite RA)
A.joint involvement | 1 day
  1 large joint (score 0) 2-10 large joints (score 1) 1-3 small joints (with or without involvement of large joints)#(score2) 4-10 small joints (with or without involvement of large joints)(score 3) 10 joints (at least 1 small joint) (score 5)
B.Serology (at least 1 test result is needed for classification) | 1 day
  Negative RF and negative ACPA (Score 0) Low-positive RF or low-positive ACPA( anticitrullinated protein antibody) (score 2) High-positive RF(rheumatoid factor) or high-positive ACPA (score 3)
C.Acute-phase reactants (at least 1 test result is needed for classification) | 1 day
  Normal CRP (C-reactive protein and normal) and normal ESR (erythrocyte sedimentation rate) (score 0) Abnormal CRP or abnormal ESR (score1)
D.Duration of symptoms | 1 day
  <6 weeks (score 0) >6 weeks (score 1)
Uromodulin measure | 1 day
  First urine sample taken in the morning

SECONDARY OUTCOMES:
CKD-EPI (Chronic Kidney Disease Epidemiology Colloboration) | 1 day
  For estimating the glomerular filtration rate
MDRD (Modification of Diet in Renal Disease) | 1 day
  For estimating the glomerular filtration rate
Urea measure | 1 day
  Fasting blood samples taken in the morning
Creatinine measure | 1 day
  Fasting blood samples taken in the morning
Sedimantation measure | 1 day
  Fasting blood samples taken in the morning
pH measure | 1 day
  First urine sample taken in the morning
Microalbuminuria measure | 1 day
  First urine sample taken in the morning

CONTACTS AND LOCATIONS:
Overall Officials: neval aksoy, MD, Study Chair — Sağlık Bilimleri Universty; lüfiye aytüre, MD, Principal Investigator — sağlık Bilimleri Universty
Locations (1):
- Istanbul saglık Bilimleri Universty Gaziosmanpaşa Egitim ve Araştırma Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided